CLINICAL TRIAL: NCT05417867
Title: Associations of Fatigue and Chemotherapy-Induced Nausea With Changes in Gut Microbiome Composition Profiles
Brief Title: Evaluating the Association Between Changes in the Gut Microbiome, Fatigue, and Chemotherapy-Induced Nausea in Early Stage Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 20-009279; NCI-2022-01231 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-05-26; First posted 2022-06-14 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Chemotherapy-Related Nausea and/or Vomiting; Early Stage Breast Carcinoma; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo collection of stool and blood samples and complete questionnaires on study.
  Interventions: Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of stool and blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This pilot study seeks to understand how changes in the bacteria composition (microbiome) of the gut may be associated with the occurrence of fatigue and chemotherapy-induced nausea (CIN) in women undergoing chemotherapy for early stage breast cancer. Patients undergoing chemotherapy may experience fatigue or nausea as a result of their treatment. Known risk factors for fatigue and CIN do not explain the differences in fatigue and CIN occurrence between patients, but changes in the functions of the gut microbiome may be related to the occurrence of fatigue and CIN. This study collects stool samples from breast cancer patients before and after chemotherapy to evaluate how changes in the microbiome may be associated with fatigue and CIN.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the feasibility of patient recruitment and retention, as well as specimen collection.

II. Estimate the effect size for changes in gut microbiome composition profiles and metabolites in stool as well as blood from time of first stool sample collection prior to chemotherapy (T1) to time of second stool sample collection after chemotherapy (T2) that are associated with the occurrence of fatigue and CIN.

III. Evaluate associations between patient reported demographic and clinical characteristics, comorbidities at T1, and changes in gastrointestinal and neuropsychological symptoms, food intake as well as exercise from T1 to T2 with the occurrence of fatigue and CIN.

OUTLINE: This is an observational study.

Patients undergo collection of stool and blood samples and complete questionnaires on study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of early stage breast cancer planning to receive moderate to highly emetogenic chemotherapy will be recruited at Mayo Clinic Health Systems including Mankato and Albert Lea; Mayo Clinic Arizona; Mayo Clinic Rochester (Minnesota); and Mayo Clinic Florida
* At least 20 years of age
* Last chemotherapy more than 3 years ago
* Scheduled to receive moderate to highly emetogenic chemotherapy with or without targeted therapies including immunotherapies

Exclusion Criteria:

* Metastatic disease
* Concurrent radiation therapy
* Concurrent antibiotic treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with a diagnosis of early stage breast cancer, planning to receive moderate to highly emetogenic chemotherapy will be recruited at Mayo Clinic Health Systems including Mankato and Albert Lea, Mayo Clinic Arizona, Mayo Clinic, Minnesota, and Mayo Clinic Florida.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of patients approached | Up to 24 months
  Assessed using descriptive statistics.
Number of patients enrolled | Up to 24 months
  Assessed using descriptive statistics.
Number of patients who completed the questionnaires at both assessments | At baseline and 3-5 days after initiation of chemotherapy
  Assessed using descriptive statistics.
Number of patients who provided stool samples at both assessments | At baseline and 3-5 days after initiation of chemotherapy
  Assessed using descriptive statistics.
Bacterial composition of stool samples | Up to study completion
  All stool samples will be processed for deoxyribonucleic acid extraction. The hypervariable regions V3 and V4 of the bacterial 16S ribosomal ribonucleic acid (rRNA) gene will be sequenced to determine bacterial composition. After quality control, 16S rRNA reads will be analyzed to determine operational taxonomic units (OTU) for T1 and T2 samples using QIIME software. Alpha (within sample) diversity and beta (between sample) diversity will be analyzed using nonmetric multidimensional scaling ordination and the effect size for changes in OTUs in gut microbiome composition profiles from T1 to T2 in patients who do and do not report fatigue or chemotherapy-induced nausea (CIN) at T2 as measured by questionnaire.
Differences in demographic between patients who do and do not report fatigue and CIN | Up to study completion
  Evaluated using parametric and non-parametric tests. The changes in gastrointestinal and neuropsychological symptoms, food intake as well as exercise from T1 to T2 associated with the occurrence of fatigue and CIN will be evaluated.
Differences in clinical characteristics between patients who do and do not report CIN | Up to study completion
  Evaluated using parametric and non-parametric tests. The changes in gastrointestinal and neuropsychological symptoms, food intake as well as exercise from T1 to T2 associated with the occurrence of CIN will be evaluated.
Differences in comorbidities between patients who do and do not report CIN | Up to study completion
  Evaluated using parametric and non-parametric tests. The changes in gastrointestinal and neuropsychological symptoms, food intake as well as exercise from T1 to T2 associated with the occurrence of CIN will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda J. Ernst, MD, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System in Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials